CLINICAL TRIAL: NCT04994886
Title: Restoring Hemodynamic Stability Using Targeted Epidural Spinal Stimulation Following Spinal Cord Injury
Acronym: STIMO HEMO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: New study in place HemON (SNCTP 000004706)
Sponsor: Jocelyne Bloch (Other)
Responsible Party: Sponsor-Investigator, Jocelyne Bloch, Professor, Neurosurgeon, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STIMO-HEMO2021
Record Dates: First submitted 2021-06-03; First posted 2021-08-06 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-02

CONDITIONS: Spinal Cord Injuries
Keywords: SCI; Spinal Cord Injury; Epidural Spinal Stimulation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Single-site, single-arm, non-blinded, non-randomized, interventional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Targeted Epidural Spinal Stimulation (Experimental): Participants will undergo a surgery for Targeted Epidural Spinal Stimulation (TESS). The neurostimulation system will be used to manage blood pressure instability.
  Patients will then proceed to one month of an intensive device configuration protocol to configure the TESS settings of their investigational device to regain hemodynamic stability. After the intensive device configuration phase, daily supervised at-home hemodynamic TESS will be tested for 5 sessions per week for two weeks. Thereafter, and up to 10 months post-implant, patients will have a minimum of 5 TESS supported at-home sessions per week and one laboratory visit per month during a long-term at-home hemodynamic TESS phase. Finally, patients will have to undergo additional testing during a configuration of additional TESS programs phase. During this phase TESS configurations for hemodynamic stability, respiratory function, trunk stability and spasticity will be tested.
  Interventions: Procedure: Device implantation

INTERVENTIONS:
Procedure: Device implantation — The intervention involves the insertion of 2 lead electrodes (Specify Surescan 5-6-5 Leads, Model 977C190 Medtronic) epidurally over the dorsal aspect of the spinal cord through 2 laminectomies and two implantable pulse generators (Intellis™ with AdaptiveStim™, Model 97715 Medtronic) in the abdomen of the participant.

SUMMARY:
The purpose of this study is to stimulate the circuits in the spinal cord that are directly responsible for hemodynamic control to restore hemodynamic stability in patients with chronic cervical or high-thoracic spinal cord injury. The ultimate objective of this feasibility study is to provide preliminary safety and efficacy measures on the ability of the hemodynamic Targeted Epidural Spinal Stimulation (TESS) to ensure the long-term management of hemodynamic instability and reduce the incidence and severity of orthostatic hypotension and autonomic dysreflexia episodes in humans with chronic cervical or high-thoracic spinal cord injury. In addition, the long-term safety and efficacy of TESS on cardiovascular health, respiratory function, spasticity, trunk stability and quality of life in patients with chronic spinal cord injury will be evaluated.

DETAILED DESCRIPTION:
The investigators hypothesize that Targeted Epidural Spinal Stimulation (TESS) foreshadows a new era in the hemodynamic management of both acute and chronic SCI. It is envisioned that TESS will become the first-line treatment for hemodynamic instability in people with chronic SCI, where vasopressor agents and compression garments will become second-line treatments behind the precise control of blood pressure achieved with TESS.

In this study, the investigators propose to investigate the preliminary safety of hemodynamic TESS to modulate pressor responses and manage blood pressure instability in 4 patients with chronic SCI located between C3 and T6 and who suffer from severe orthostatic hypotension.

The study intervention consists of 8 phases preceded by pre-screening:

* Screening and enrolment
* Baseline and pre-implantation assessments
* Surgery
* Intensive TESS Configuration phase
* Daily supervised at-home TESS phase
* Long-term at-home phase
* Configuration of additional TESS programs phase
* End of study

Measures will be performed before surgical intervention and at regular intervals during the study.

The study will take place at the CHUV (Lausanne, Switzerland). A total of 4 participants will be enrolled in the study and implanted with two lead electrodes (Specify Surescan 5-6-5 Leads, Model 977C190 Medtronic) and two implantable pulse generators (Intellis™ with AdaptiveStim™, Model 97715 Medtronic). All participants will undergo the same treatment and procedures. The total duration of the study will be approximately 2 months (up to 10 months/participant).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years old
* Able to undergo the informed consent/assent process
* Radiologically confirmed spinal cord injury
* Spinal cord injury between C3 and T6
* Classified with AIS A or B Spinal cord injury
* Stable medical, physical and psychological condition as considered by Investigators
* Greater than 1 year since initial injury and at least 6 months from any required spinal instrumentation
* Confirmed orthostatic hypotension and autonomic dysreflexia
* Willing to attend all scheduled appointments

Exclusion Criteria:

* Patients in an emergency situation
* Diseases and conditions that would increase the morbidity and mortality of spinal cord injury surgery
* The inability to withhold antiplatelet/anticoagulation agents perioperatively
* History of myocardial infarction or cerebrovascular event
* Other conditions that would make the subject unable to participate in testing in the judgment of the investigators
* Current and anticipated need for opioid pain medications or pain that would prevent full participation in the rehabilitation program in the judgement of the investigators
* Clinically significant mental illness in the judgment of the investigators
* Botulinum toxin injections in the previous 6 months
* Presence of significant pressure ulcers
* Recurrent urinary tract infection refractory to antibiotics
* Current pregnancy
* Current breastfeeding
* Known or suspected drug or alcohol abuse
* Unhealed spinal fractures
* Presence of indwelling baclofen or insulin pump

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Occurrence of Adverse Events and Serious Adverse Events that are deemed related or possibly related to the study procedure or to the study investigational system, from implant surgery until the end of study. | From implantation through study completion, an average of 7 months
  Investigate the preliminary safety of hemodynamic targeted epidural spinal stimulation (TESS) to modulate pressor responses and manage blood pressure instability in patients with chronic SCI located between C3 and T6 and who suffer from severe orthostatic hypotension (n=4).

SECONDARY OUTCOMES:
ISNCSCI (International Standards for Neurological Classification of Spinal Cord Injury) | At baseline and during the rehabilitation phase, an average of 7 months
  Clinical examination used to assess the motor and sensory impairment and severity of a spinal cord injury.
Spasticity clinical exam using the Modified Ashworth Scale (MAS) | At baseline and during the rehabilitation phase, an average of 7 months
  Patient's limb spasticity levels (5-point nominal scale) are assessed by rating the resistance of a muscle to a passive range of motion about a single joint. Scores range from 0 to 4 with higher scores indicating higher spasticity.
Spasticity isokinetic quantification | At baseline and during the rehabilitation phase, an average of 7 months
  A dynamometer (Cybex) is used to evaluate the effect of stimulation on spasticity of the hip, knee and ankle. An extension and flexion movement is performed around each joint (dynamometer in isokinetic mode).
Spasticity isokinetic quantification | At baseline and during the rehabilitation phase, an average of 7 months
  An extension and flexion movement is performed around each joint. EMG data is recorded through each movement.
Trunk stability | At baseline and during the rehabilitation phase, an average of 7 months
  The patient is asked to perform a systematic set of reaching movements while seated freely (without a back-rest). Additionally, the patient is asked to perform a set of movements deemed functionally relevant, for example reaching for an object behind them or picking up an object from the ground. Each movement is repeated and EMG data can be acquired.
Respiratory function evaluation | At baseline and during the rehabilitation phase, an average of 7 months
  The respiratory function is evaluated using a spirometer. Volume is recorded.
Respiratory function evaluation | At baseline and during the rehabilitation phase, an average of 7 months
  The respiratory function is evaluated using a spirometer. Flow is recorded.
Orthostatic head-up tilt test | At baseline and during the rehabilitation phase, an average of 7 months
  Patients begin by resting in the supine position during which a baseline recording is performed. Thereafter, patients will be passively moved to upright position using the tilt-table. Between each experimental condition, the patient will be moved back in supine position to return to baseline. Beat-to-beat blood pressure will be monitored.
Autonomic Dysfunction Following Spinal cord injury (ADFSCI) | At baseline and monthly during the rehabilitation phase, an average of 7 months
  The ADFSCI questionnaire is a 24-item self-reported questionnaire. The questionnaire consists of demographics, medications, frequency/severity of symptoms during AD and hypotensive events. Higher scores indicate more severe and more frequent symptoms during AD and hypotensive events.
Quality of Life questionnaire WHOQOL-BREF | At baseline and monthly during the rehabilitation phase, an average of 7 months
  The WHOQOL-BREF is a questionnaire used to assess the quality of life. Scores are converted to range between 4-20 or 0-100 and are scaled in a positive direction: higher scores denote higher quality of life.
Completion of a Daily Stimulation Log (DSL) by the patient | From daily at-home supervised used until the end of the study, an average of 5 months
  The patient will be asked to self-report the use of TESS during the at-home phases. This information will be used to evaluate hemodynamic TESS-supported at-home stimulation sessions and characterize the use of the investigational system at home.

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyne Bloch, MD, Principal Investigator — CHUV
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson KD. Targeting recovery: priorities of the spinal cord-injured population. J Neurotrauma. 2004 Oct;21(10):1371-83. doi: 10.1089/neu.2004.21.1371. PMID 15672628
- [Background] Cragg JJ, Noonan VK, Krassioukov A, Borisoff J. Cardiovascular disease and spinal cord injury: results from a national population health survey. Neurology. 2013 Aug 20;81(8):723-8. doi: 10.1212/WNL.0b013e3182a1aa68. Epub 2013 Jul 24. PMID 23884034
- [Background] Illman A, Stiller K, Williams M. The prevalence of orthostatic hypotension during physiotherapy treatment in patients with an acute spinal cord injury. Spinal Cord. 2000 Dec;38(12):741-7. doi: 10.1038/sj.sc.3101089. PMID 11175374
- [Background] Phillips AA, Krassioukov AV. Contemporary Cardiovascular Concerns after Spinal Cord Injury: Mechanisms, Maladaptations, and Management. J Neurotrauma. 2015 Dec 15;32(24):1927-42. doi: 10.1089/neu.2015.3903. Epub 2015 Sep 1. PMID 25962761
- [Background] Phillips AA, Krassioukov AV, Ainslie PN, Warburton DE. Perturbed and spontaneous regional cerebral blood flow responses to changes in blood pressure after high-level spinal cord injury: the effect of midodrine. J Appl Physiol (1985). 2014 Mar 15;116(6):645-53. doi: 10.1152/japplphysiol.01090.2013. Epub 2014 Jan 16. PMID 24436297
- [Background] Phillips AA, Warburton DE, Ainslie PN, Krassioukov AV. Regional neurovascular coupling and cognitive performance in those with low blood pressure secondary to high-level spinal cord injury: improved by alpha-1 agonist midodrine hydrochloride. J Cereb Blood Flow Metab. 2014 May;34(5):794-801. doi: 10.1038/jcbfm.2014.3. Epub 2014 Jan 29. PMID 24473484
- [Background] Phillips AA, Elliott SL, Zheng MM, Krassioukov AV. Selective alpha adrenergic antagonist reduces severity of transient hypertension during sexual stimulation after spinal cord injury. J Neurotrauma. 2015 Mar 15;32(6):392-6. doi: 10.1089/neu.2014.3590. Epub 2014 Dec 5. PMID 25093677
- [Background] Krassioukov A, Eng JJ, Warburton DE, Teasell R; Spinal Cord Injury Rehabilitation Evidence Research Team. A systematic review of the management of orthostatic hypotension after spinal cord injury. Arch Phys Med Rehabil. 2009 May;90(5):876-85. doi: 10.1016/j.apmr.2009.01.009. PMID 19406310
- [Background] Squair JW, Phillips AA, Harmon M, Krassioukov AV. Emergency management of autonomic dysreflexia with neurologic complications. CMAJ. 2016 Oct 18;188(15):1100-1103. doi: 10.1503/cmaj.151311. Epub 2016 May 24. No abstract available. PMID 27221275
- [Background] Phillips AA, Krassioukov AV, Ainslie PN, Warburton DE. Baroreflex function after spinal cord injury. J Neurotrauma. 2012 Oct 10;29(15):2431-45. doi: 10.1089/neu.2012.2507. Epub 2012 Sep 20. PMID 22897489
- [Background] Courtine G, Gerasimenko Y, van den Brand R, Yew A, Musienko P, Zhong H, Song B, Ao Y, Ichiyama RM, Lavrov I, Roy RR, Sofroniew MV, Edgerton VR. Transformation of nonfunctional spinal circuits into functional states after the loss of brain input. Nat Neurosci. 2009 Oct;12(10):1333-42. doi: 10.1038/nn.2401. Epub 2009 Sep 20. PMID 19767747
- [Background] Wagner FB, Mignardot JB, Le Goff-Mignardot CG, Demesmaeker R, Komi S, Capogrosso M, Rowald A, Seanez I, Caban M, Pirondini E, Vat M, McCracken LA, Heimgartner R, Fodor I, Watrin A, Seguin P, Paoles E, Van Den Keybus K, Eberle G, Schurch B, Pralong E, Becce F, Prior J, Buse N, Buschman R, Neufeld E, Kuster N, Carda S, von Zitzewitz J, Delattre V, Denison T, Lambert H, Minassian K, Bloch J, Courtine G. Targeted neurotechnology restores walking in humans with spinal cord injury. Nature. 2018 Nov;563(7729):65-71. doi: 10.1038/s41586-018-0649-2. Epub 2018 Oct 31. PMID 30382197
- [Background] Squair JW, Gautier M, Mahe L, Soriano JE, Rowald A, Bichat A, Cho N, Anderson MA, James ND, Gandar J, Incognito AV, Schiavone G, Sarafis ZK, Laskaratos A, Bartholdi K, Demesmaeker R, Komi S, Moerman C, Vaseghi B, Scott B, Rosentreter R, Kathe C, Ravier J, McCracken L, Kang X, Vachicouras N, Fallegger F, Jelescu I, Cheng Y, Li Q, Buschman R, Buse N, Denison T, Dukelow S, Charbonneau R, Rigby I, Boyd SK, Millar PJ, Moraud EM, Capogrosso M, Wagner FB, Barraud Q, Bezard E, Lacour SP, Bloch J, Courtine G, Phillips AA. Neuroprosthetic baroreflex controls haemodynamics after spinal cord injury. Nature. 2021 Feb;590(7845):308-314. doi: 10.1038/s41586-020-03180-w. Epub 2021 Jan 27. PMID 33505019
- [Background] Legg Ditterline BE, Aslan SC, Wang S, Ugiliweneza B, Hirsch GA, Wecht JM, Harkema S. Restoration of autonomic cardiovascular regulation in spinal cord injury with epidural stimulation: a case series. Clin Auton Res. 2021 Apr;31(2):317-320. doi: 10.1007/s10286-020-00693-2. Epub 2020 May 13. No abstract available. PMID 32405661
- [Background] Harkema SJ, Legg Ditterline B, Wang S, Aslan S, Angeli CA, Ovechkin A, Hirsch GA. Epidural Spinal Cord Stimulation Training and Sustained Recovery of Cardiovascular Function in Individuals With Chronic Cervical Spinal Cord Injury. JAMA Neurol. 2018 Dec 1;75(12):1569-1571. doi: 10.1001/jamaneurol.2018.2617. PMID 30242310
- [Background] Aslan SC, Legg Ditterline BE, Park MC, Angeli CA, Rejc E, Chen Y, Ovechkin AV, Krassioukov A, Harkema SJ. Epidural Spinal Cord Stimulation of Lumbosacral Networks Modulates Arterial Blood Pressure in Individuals With Spinal Cord Injury-Induced Cardiovascular Deficits. Front Physiol. 2018 May 18;9:565. doi: 10.3389/fphys.2018.00565. eCollection 2018. PMID 29867586
- [Background] Harkema SJ, Wang S, Angeli CA, Chen Y, Boakye M, Ugiliweneza B, Hirsch GA. Normalization of Blood Pressure With Spinal Cord Epidural Stimulation After Severe Spinal Cord Injury. Front Hum Neurosci. 2018 Mar 8;12:83. doi: 10.3389/fnhum.2018.00083. eCollection 2018. PMID 29568266